CLINICAL TRIAL: NCT07032610
Title: Long-term Immunogenicity of Lived-attenuated Hepatitis A Virus Vaccine Among Healthy Thai Children and Adolescents
Brief Title: Long-term Immunogenicity of L-HAV Vaccine Among Healthy Thai Children and Adolescents
Status: Not yet recruiting | Type: Observational
Sponsor: Chiang Mai University (Other)
Collaborators: Faculty of Medicine, Chiang Mai University (Unknown)
Responsible Party: Principal Investigator, Tavitiya Sudjaritruk, Associate Professor, Chiang Mai University
Other Study IDs: PED-2568-0420
Record Dates: First submitted 2025-06-16; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis A; Hepatitis A Virus; Vaccine-Preventable Diseases
Keywords: Live-attenuated hepatitis A vaccine; Immunogenicity; Seropositive rate
MeSH Terms: conditions — Hepatitis A; Hepatitis; Vaccine-Preventable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatitis A virus (HAV) remains a common infection among Thai children. Two types of HAV vaccines are available in Thailand: an inactivated vaccine (I-HAV, administered in two doses 6 months apart) and a live-attenuated vaccine (L-HAV, administered as a single dose). However, neither vaccine is currently included in Thailand's Expanded Programme on Immunization (EPI). In 2024, a randomized, active-controlled, open-label, non-inferiority trial was conducted to compare the immunogenicity and safety of the two-dose I-HAV with the single-dose L-HAV in healthy Thai children and adolescents aged 18 months to 18 years. This study aims to evaluate the long-term seropositive rate and immunogenicity of anti-HAV antibodies in this population following a single dose of L-HAV.

DETAILED DESCRIPTION:
Hepatitis A virus (HAV) infection remains one of the most common causes of viral hepatitis among children and adolescents in developing countries, including Thailand. The virus is primarily transmitted through the ingestion of contaminated food or water, or through direct contact with an infected person. HAV typically causes acute hepatitis, ranging from mild illness to severe fulminant hepatitis (acute liver failure), but it does not lead to chronic liver disease. Vaccination is a highly effective strategy to prevent HAV infection and its serious complications.

Currently, two types of HAV vaccines are available in Thailand: (1) the inactivated HAV vaccine (I-HAV), which is administered in two doses six months apart and is approved for use in children aged 12 months and older; and (2) the live-attenuated HAV vaccine (L-HAV), administered as a single dose and approved for children aged 18 months and older. However, neither vaccine has been included in Thailand's Expanded Programme on Immunization (EPI), resulting in suboptimal vaccination coverage across the country.

In 2024, the investigators conducted a randomized, active-controlled, open-label, non-inferiority trial to compare the immunogenicity and safety of the two-dose I-HAV regimen with the single-dose L-HAV in healthy Thai children and adolescents aged 18 months to 18 years. The present study aims to assess the long-term seropositive rate and immunogenicity of anti-HAV antibodies among these participants following a single dose of L-HAV.

ELIGIBILITY:
Inclusion Criteria:

* Thai children and adolescents who previously participated in the previous RCT study
* Previously randomized to receive one dose of L-HAV vaccine within the past 1 year (+/- 3 months)
* Participants and/or caregivers gives written inform consent/assent form

Exclusion Criteria:

* History of acute illness within 4 weeks prior to study enrollment
* Has a history of illness or a diagnosis consistent with hepatitis A after receiving the live attenuated hepatitis A vaccine as part of participation in a previous research study
* Has a history of receiving any additional hepatitis A vaccine after participating in the previous research study
* Presence of fever (body temperature ≥38.0°C), jaundice, or yellowing of the eyes within 4 weeks prior to study enrollment
* Have any condition that, in the opinion of the site investigator, would compromise the subject's ability to participate in the study

Ages: 18 Months to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy Thai children and adolescents age 18 months to 20 years who received a single dose of L-HAV vaccine in the previous RCT study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-22 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Anti-HAV seropositivity rate | 1 year after L-HAV vaccination
  Anti-HAV seropositivity rate following a single L-HAV vaccine
Anti-HAV antibody level | 1 year after L-HAV vaccination
  Geometric mean concentration (GMC) of anti-HAV antibodies following a single L-HAV vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Tavitiya Sudjaritruk, MD, PhD, Study Chair — Department of Pediatrics, Faculty of Medicine, Chiang Mai University; Natchaya Kunanitthaworn, MD, Principal Investigator — Department of Pediatrics, Faculty of Medicine, Chiang Mai University
Locations (1):
- Department of Pediatrics, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available to other researchers for this study.

REFERENCES:
- [Background] Ma F, Yang J, Kang G, Sun Q, Lu P, Zhao Y, Wang Z, Luo J, Wang Z. Comparison of the safety and immunogenicity of live attenuated and inactivated hepatitis A vaccine in healthy Chinese children aged 18 months to 16 years: results from a randomized, parallel controlled, phase IV study. Clin Microbiol Infect. 2016 Sep;22(9):811.e9-811.e15. doi: 10.1016/j.cmi.2016.06.004. Epub 2016 Jun 23. PMID 27345175
- [Background] Liu XE, Wushouer F, Gou A, Kuerban M, Li X, Sun Y, Zhang J, Liu Y, Li J, Zhuang H. Comparison of immunogenicity between inactivated and live attenuated hepatitis A vaccines: a single-blind, randomized, parallel-group clinical trial among children in Xinjiang Uighur Autonomous Region, China. Hum Vaccin Immunother. 2013 Jul;9(7):1460-5. doi: 10.4161/hv.24366. Epub 2013 Apr 9. PMID 23571173
- [Result] Kunanitthaworn N, Mueangmo O, Saheng J, Wongjak W, Lertsiriladakul T, Chaito T, Nantarat P, Sudjaritruk T. Seroprevalence of hepatitis A virus antibodies among children and adolescents living in Northern Thailand: an implication for hepatitis A immunization. Sci Rep. 2023 Oct 13;13(1):17432. doi: 10.1038/s41598-023-44643-0. PMID 37833325